CLINICAL TRIAL: NCT04792892
Title: ANCA II - Quality of Life and Functional Outcome in Patients With Anal Cancer
Acronym: ANCAII
Status: Recruiting | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Eva Angenete, Professor, Sahlgrenska University Hospital
Other Study IDs: ANCA II
Record Dates: First submitted 2021-03-10; First posted 2021-03-11 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Anal Cancer
MeSH Terms: conditions — Anus Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with a new diagnosis of anal cancer: All patients identified at our national tumour board will be offered to participate
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Patients will be answering questionnaires at 0, 3, 12, 36, 60 and 120 months

SUMMARY:
Anal cancer is a rare disease, but the incidence is rising. About 200 patients will get this type of cancer yearly in Sweden. Curative treatment includes chemotherapy and radiotherapy. The prognosis is good, but some patients will have recurrent or persistent disease after concluded chemo-radiotherapy and will then be offered salvage surgery. Some patients develop distant metastases that can be treated with good results.

The aim of this study is to identify and describe functional outcome in patients diagnosed with anal cancer. We will study patients from diagnosis, try to identify early toxicity to treatment and then identify long-term morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Anal squamous carcinoma diagnosed within the last 2 months

Exclusion Criteria:

-No informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed anal cancer
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2035-04-01 (Estimated)

PRIMARY OUTCOMES:
QoL | 3 months after diagnosis
  Health related QoL at
Urinary function | 3 months after diagnosis
  Evaluate urinary dysfunction
Bowel function | 3 months after diagnosis
  Evaluate bowelfunction
Sexual function | 3 months after diagnosis
  Evaluate sexual function
Toxicity related to treatment | 3 months after diagnosis
  Number of patients with severe toxicity from the chemoradiotherapy

SECONDARY OUTCOMES:
QoL | 12 months after diagnosis
  QoL measured on a 7 point likert scale at 12 months
Urinary function | 12 months after diagnosis
  Urinary dysfuntion measured as incontinence at 12 months
Bowel function | 12 months after diagnosis
  Bowel dysfunction measured at 12 months
Sexual function | 12 months after diagnosis
  Sexual dysfunction measured at 12 months
QoL | 3 years after diagnosis
  QoL measured on a 7 point likert scale at 3 years
Urinary function | 3 years after diagnosis
  Urinary function at 3 years
Bowel funcction | 3 years after diagnosis
  Bowel dysfunction at 3 years
Sexual function | 3 years after diagnosis
  Sexual dysfunction at 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Surgery, Sahlgrenska University Hospital/Ostra, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided